CLINICAL TRIAL: NCT02475967
Title: eEduHeart I: a Multi-center Randomized, Controlled Trial Investigating the Effectiveness of a Cardiac Web-based eLearning Platform
Brief Title: Study Assessing the Effectiveness of a Cardiac Web-based eLearning Platform
Acronym: eEduHeart I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PDEN-IFRE 01
Record Dates: First submitted 2015-06-10; First posted 2015-06-19 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
Keywords: E-Learning; coronary artery disease; telerehabilitation; e-health
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group patients have access to the eLearning platform in addition to conventional cardiac care.
  Interventions: Other: Intervention group
- Control group (Active Comparator): The control group patients receive conventional cardiac care alone.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — The intervention group patients have access to the eLearning platform in addition to conventional cardiac care.The content of platform will be gathered from a multidisciplinary input of both medics (e.g. cardiologists) and paramedics (e.g. psychologists). Patients will also contribute to platform content.
  Arms: Intervention group
Other: Control group — The control group patients receive conventional cardiac care alone.
  Arms: Control group

SUMMARY:
In the trial cardiac patients will be provided with unrestricted access to the web-based eLearing platform for a one-month period.

DETAILED DESCRIPTION:
Patients participating in the trial will be provided with a cardiac web-based eLearning platform for one month during study period. The medical content of the packages will be gathered from a multidisciplinary input of both medics (e.g. cardiologists) and paramedics (e.g. psychologists).

E-Learning packages type I: videos with information from caregivers. In these videos, medics and paramedics are interviewed to highlight the etiology, pathophysiology and treatment of coronary artery disease; the associated comorbidities and the ways to prevent recurrence.

E-Learning packages type II: videos in which patients are interviewed. Patients can help each other to adhere to their treatment plan, by sharing stories from their own experience about their illness and the rehabilitation afterwards. Short clips of maximum 2 minutes will be provided to study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from coronary artery disease for which they are treated conservatively, with a percutaneous coronary intervention or with coronary artery bypass grafting

Exclusion Criteria:

* Patients with dementia or cognitive impairment not being able to sufficiently understand the E-Learning packages content
* (Foreign) patients unable to speak Dutch, thereby not being able to understand the content of the E-Learning packages
* Patients with advanced visual and/or auditory impairments, hindering them to adequately understand the E-earning packages
* Patients participating in another trial during the Pilot study period
* Patients refusing to provide signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 3 months
  Health-related quality of life, assessed by HeartQol

SECONDARY OUTCOMES:
Adherence to the E-learning packages | 3 months
  Adherence to the E-learning packages as assessed by the number of logs and the cumulative log time on the E-learning platform per patient.
Effectiveness of E-learning packages | 3 months
  Effectiveness of intervention in improving patients' knowledge of cardiac diseases as assessed by questionnaire scores.
User experience of eLearning platform | 3 months
  Asses user experience of eLearning platform by User Experience Questionnaire (UEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ines Frederix, drs., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - ZOL, Genk
  - Jessa Ziekenhuis, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided